CLINICAL TRIAL: NCT04353336
Title: Clinical Study Evaluating the Efficacy of Chloroquine or Hydroxychloroquine in COVID-19 Treatment
Brief Title: Efficacay of Chloroquine or Hydroxychloroquine in COVID-19 Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: chloroquine covid
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: COVID-19; Coronavirus Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Chloroquine; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chloroquine or Hydroxychloroquine (Experimental): Chloroquine or Hydroxychloroquine with standard of care treatment.
  Interventions: Drug: Chloroquine or Hydroxychloroquine
- No intervention (No Intervention): standard of care treatment alone.

INTERVENTIONS:
Drug: Chloroquine or Hydroxychloroquine — Chloroquine or Hydroxychloroquine
  Other Names: alexoquine, chloroquine, Hydroquine
  Arms: Chloroquine or Hydroxychloroquine

SUMMARY:
Chloroquine or hydroxychloroquine in COVID-19 treatment

DETAILED DESCRIPTION:
Clinical Study Evaluating the Efficacy of Chloroquine or hydroxychloroquine in COVID-19 treatment

ELIGIBILITY:
Inclusion Criteria:

* Covid 19 patients

Exclusion Criteria:

* Allergy or contraindication to the drug
* Pregnant or lactating
* Patients with cardiac problems

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with cure or death | 1 month
  the number of patients with cure or death

CONTACTS AND LOCATIONS:
Overall Officials: sherief Abd-Elsalam, Ass. Prof., Principal Investigator — Tanta University - Faculty of Medicine
Locations (1):
- Tanta University, Assiut University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No